CLINICAL TRIAL: NCT03167762
Title: Fluorescence and Thermal Imaging of the Skin Before and During Photodynamic Therapy
Brief Title: Photographing the Skin During Photodynamic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17/WS/0055
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Basal Cell Carcinoma; Bowen's Disease
MeSH Terms: conditions — Carcinoma, Basal Cell; Bowen's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental)
  Interventions: Device: Fluorescence and thermal imaging

INTERVENTIONS:
Device: Fluorescence and thermal imaging — Two cameras used to take images of the skin. One, to measure the fluorescence from the photosensitiser, and the second to measure the surface temperature of the skin

SUMMARY:
Photodynamic therapy (PDT) is used to treat some types of sun-damaged skin and low-grade forms of growths. A cream is applied to the skin, and the chemical in this cream is absorbed in to the skin and converted in to a 'photosensitiser'. This photosensitiser is fluorescent, meaning that it produces red light when blue light is shone on it. By measuring how much light is given off with a camera, the investigators can determine how much photosensitiser is present in the skin. Also, it is thought that more of the chemical is converted to the active photosensitiser if the skin is warmer, so the investigators plan to measure the temperature of the skin using a thermal camera. Light is shone on to the skin and this activates the photosensitiser, treating the problem area and leaving healthy skin intact. This research will increase the investigators understanding of how PDT works, and may help the investigators to improve treatment regimens so that they can be made more effective and better tolerated

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients presenting with superficial BCC or Bowen's disease (one or two lesions and diagnosed either clinically or histologically and untreated or having had no treatment for 4 months or longer) 2. Adult males and females, >18 years only 3. Capable of giving informed consent 4. Able to understand and adhere to protocol requirements

Exclusion Criteria:

* 1. Patients skin lesions have had previous treatment in the last 4 months 2. Unable to give informed consent 3. Known allergy to Metvix® 4. Known to have a light sensitive disorder 5. Pregnant, breastfeeding or planning to conceive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Is there a correlation between body site temperature and degree of fluorescence prior to and/or during PDT | 12months
  Body site temperature is measured before and during PDT (in degrees Celsius) as is fluorescence signal (in arbitrary fluorescence units). These are compared for each time point in the treatment for each patient.

SECONDARY OUTCOMES:
Is there a correlation between temperature and/or fluorescence and treatment outcome | 12months
  Following from Outcome 1, these data for each patient will be compared with the clinical outcome (determined visually by Dermatologist) at 3 and 12 months, to see if there is a correlation between either measurements and clinical outcome.
How does the spatial distribution of fluorescence and temperature change prior to and during PDT | 12months
  Fluorescence and thermal cameras record field of view data, so the investigators can investigate how the fluorescence and thermal distribution in the lesions changes during treatment.
Pain measured immediately after irradiation | 12months
  Pain (visual analogue scale 1-10 cm-1) is measured after treatment, and the investigators will check for correlations between this properties and the fluorescence and thermal readings for each patient.
phototoxicity (inflammation) measured immediately after irradiation | 12months
  inflammation (measured visually by a Dermatologist) is measured after treatment, and the investigators will check for correlations between this property and the fluorescence and thermal readings for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Ninewells Hopsital, Dundee, Tayside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morton CA, McKenna KE, Rhodes LE; British Association of Dermatologists Therapy Guidelines and Audit Subcommittee and the British Photodermatology Group. Guidelines for topical photodynamic therapy: update. Br J Dermatol. 2008 Dec;159(6):1245-66. doi: 10.1111/j.1365-2133.2008.08882.x. Epub 2008 Oct 13. PMID 18945319
- [Background] Morton CA, Szeimies RM, Sidoroff A, Braathen LR. European guidelines for topical photodynamic therapy part 1: treatment delivery and current indications - actinic keratoses, Bowen's disease, basal cell carcinoma. J Eur Acad Dermatol Venereol. 2013 May;27(5):536-44. doi: 10.1111/jdv.12031. Epub 2012 Nov 26. PMID 23181594
- [Background] Valentine RM, Ibbotson SH, Wood K, Brown CT, Moseley H. Modelling fluorescence in clinical photodynamic therapy. Photochem Photobiol Sci. 2013 Jan;12(1):203-13. doi: 10.1039/c2pp25271f. PMID 23128146
- [Background] Mamalis A, Koo E, Sckisel GD, Siegel DM, Jagdeo J. Temperature-dependent impact of thermal aminolaevulinic acid photodynamic therapy on apoptosis and reactive oxygen species generation in human dermal fibroblasts. Br J Dermatol. 2016 Sep;175(3):512-9. doi: 10.1111/bjd.14509. Epub 2016 Jul 24. PMID 26931503
- [Result] Kulyk O, Ibbotson SH, Moseley H, Valentine RM, Samuel ID. Development of a handheld fluorescence imaging device to investigate the characteristics of protoporphyrin IX fluorescence in healthy and diseased skin. Photodiagnosis Photodyn Ther. 2015 Dec;12(4):630-9. doi: 10.1016/j.pdpdt.2015.10.002. Epub 2015 Oct 20. PMID 26467274